CLINICAL TRIAL: NCT06187142
Title: Mobile Phone-Based Smoking-Cessation Intervention for Chronic Patients: a Sequential, Multiple Assignment, Randomized Trial (SMART)
Brief Title: Mobile Phone-Based Smoking-Cessation Intervention for Chronic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: mCessation in Chronic Patients
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Chronic patients; SMART design
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Group PCS, subgroup PCS-1+PCS-2+PCS-3) (Experimental): Personalized Chat Support (PCS) + Multi-component Optional Support (MOS) + 5A's / 5R's advice + health warning leaflet +Self-help booklet
  Interventions: Behavioral: Initial phase: Personalized Chat Support (PCS); Behavioral: Second phase: Multi-component Optional Support (MOS); Behavioral: 5A's / 5R's advice; Behavioral: health warning leaflet; Behavioral: Self-help booklet
- Control Group (Group GCS, subgroup GCS-1+GCS-2+GCS-3) (Experimental): Group Chat Support (GCS) + Personalized Chat Support (PCS) + 5A's / 5R's advice + health warning leaflet +Self-help booklet
  Interventions: Behavioral: Initial phase: Group Chat Support (GCS); Behavioral: Second phase: Personalized Chat Support (PCS); Behavioral: 5A's / 5R's advice; Behavioral: health warning leaflet; Behavioral: Self-help booklet

INTERVENTIONS:
Behavioral: Initial phase: Personalized Chat Support (PCS) — Participants will receive three months of personalized chat support through WeChat. A total of 24 pre-set messages will be sent with the schedule of 3 times a week for 2 weeks, twice a week for the next 8 weeks and once a week for the last 2 weeks. These messages cover generic information about the benefits of quitting, methods to avoid/ manage craving or withdrawal symptoms, and hazards of smoking for chronic diseases experienced by different participants. Counsellors will respond to the participants' messages instantly. At the end of the initial phase (1-month), complete responders (quitters) will continue to receive PCS (subgroup PCS-1). Incomplete responders (smokers) will be randomly assigned to continue PCS (subgroup PCS-2) or receive PCS and MOS (subgroup PCS-3).
  Arms: Intervention Group (Group PCS, subgroup PCS-1+PCS-2+PCS-3)
Behavioral: Second phase: Multi-component Optional Support (MOS) — For incomplete responders (subgroup PCS-3) randomized to MOS, the available intervention options include phone counseling, family/peer support group and financial incentive for nicotine replacement therapy. Participants will be guided by cessation counsellors at 1-month follow-up to choose any combination of MOS based on their prefer choice or combination of MOS. If MOS participants cannot be followed up at 1-month, they will continue PCS by default.
  Arms: Intervention Group (Group PCS, subgroup PCS-1+PCS-2+PCS-3)
Behavioral: Initial phase: Group Chat Support (GCS) — Participant will receive three months of group chat support through WeChat. In this group, participants can send 'No Smoking' and the smart quit-smoking assistant will record it. A smoking cessation clinic doctor in the group will respond to participants' questions about smoking cessation. At the end of the initial phase (1-month), complete responders (quitters) will continue to receive GCS (subgroup GCS-1). Incomplete responders (smokers) will be randomly assigned to continue GCS (subgroup GCS-2) or receive GCS and PCS (subgroup GCS-3).
  Arms: Control Group (Group GCS, subgroup GCS-1+GCS-2+GCS-3)
Behavioral: Second phase: Personalized Chat Support (PCS) — For incomplete responders (subgroup GCS-3) randomized to PCS, participants will receive the same intervention as Group PCS delivered at the initial stage. Participants will receive two months of personalized messages through WeChat. Please refer to Intervention Group 'Initial phase: Personalized Chat Support (PCS) for details.
  Arms: Control Group (Group GCS, subgroup GCS-1+GCS-2+GCS-3)
Behavioral: 5A's / 5R's advice — 5A's (Ask, Advise, Assess, Assist, Arrange) for smokers who are ready to quit, and 5R's (relevance, risks, rewards, roadblocks, and repetition) for smokers who are not ready to quit.
Behavioral: health warning leaflet — The contents of the leaflet include the absolute risk of smoking, diseases caused by active and second-hand smoking, horrible pictorial warnings of the health consequences of active and second-hand smoking, and the benefits of quitting.
Behavioral: Self-help booklet — The contents include information about the benefits of quitting, methods to quit, how to handle withdrawal symptoms, misperceptions of quitting, etc.

SUMMARY:
The study aims to facilitate mobile phone-based cessation support for chronic patients using a sequential multiple assignment randomized trial (SMART) , and combines different effective treatments to enhance engagement and determine the most effective adaptive interventions.

DETAILED DESCRIPTION:
Noncommunicable diseases (NCDs) , also known as chronic diseases, affect of a large of number of people and cause 41 million death each year, equivalent to 74% of globally mortality. In China, NCDs have caused 86% of deaths in the past three decades.

Tobacco use is a type of modifiable behavioural risk factor for the development of noncommunicable disease and death. It not only increases the risk of developing NCDs, but also exacerbates their severity and complications. Tobacco causes over 8 million deaths annually. China has the world's largest population of smokers, more than 300 million. Tobacco related deaths in China are 1 million per year. Smoking cessation is one of the most effective and cost-efficient measures for the prevention and control of NCDs. It can reduce the morbidity and mortality rates of NCDs and improve the health and quality of life of patients.

Meanwhile, among current smokers in China, the prevalence of tobacco dependence was 49.7%, smoking cessation services are extremely limited in China, with only 366 clinics nationwide. For smokers with NCDs, hospitalization or outpatient treatment due to health problems can be a 'teachable moment' for quit smoking. Most physicians are unable to provide comprehensive cessation advice due to time and resource constraints, and chronic patients face many relapse triggers after leaving the hospital. Therefore, it is necessary to implement staged and personalized smoking cessation interventions for chronic patients.

To facilitate smoking cessation among chronic patients, we propose to use a sequential multiple assignment randomized trial (SMART) design. This adaptive approach is a concept of stepped treatment that aims to address the unmet needs of chronic patients and enhance smoking cessation outcomes.

The study aims to facilitate mobile phone-based cessation support for chronic patients using a sequential multiple assignment randomized trial (SMART) , and combines different effective treatments to enhance engagement and determine the most effective adaptive interventions.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or above, reside in Zhuhai for next 6 months;
2. smoke at least 1 cigarette or use e-cigarettes daily;
3. having a smartphone and a WeChat account, being able to use WeChat skillfully;
4. having a diagnosis of at least one chronic disease related to smoking;
5. intent to quit / reduce smoking.

Exclusion Criteria:

1. smokers who have communication barrier (either physically or cognitively)
2. having participation in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Participation rate of eligible smokers (Feasibility) | Baseline
  The percentage of eligible smokers who agree to participate in the intervention

SECONDARY OUTCOMES:
Validated and self-reported abstinence of PCS vs. GCS | 3- and 6-month follow-up
  PCS (subgroup 1+2+3) vs. GCS(subgroup 1+2+3) on validated abstinence (salivary cotinine < 10 ng/ml) and self-reported abstinence.
Validated and self-reported abstinence of PCS-3 vs. GCS-2 | 3- and 6-month follow-up
  PCS-3 (add MOS) vs. GCS-2 (participants who are still smoking with 1-month) on validated abstinence (salivary cotinine < 10 ng/ml) and self-reported abstinence.
Validated and self-reported abstinence of PCS-3 vs. PCS-2 | 3- and 6-month follow-up
  PCS-3 (add MOS) vs. PCS-2 (participants who are still smoking with 1-month) on validated abstinence (salivary cotinine < 10 ng/ml) and self-reported abstinence.
Validated and self-reported abstinence of GCS-3 vs. GCS-2 | 3- and 6-month follow-up
  GCS-3 (add PCS) vs. GCS-2 (participants who are still smoking with 1-month) on validated abstinence (salivary cotinine < 10 ng/ml) and self-reported abstinence.
Validated and self-reported abstinence of PCS-1+2 vs. GCS-1+2 | 3- and 6-month follow-up
  PCS-1+2 vs. GCS-1+2 on validated abstinence (salivary cotinine < 10 ng/ml) and self-reported abstinence.
Smoking reduction rate | 3- and 6-months follow-up
  Rate of smoking reduction by at least half of baseline amount in different groups.
Engagement in PCS / GCS intervention | 3- and 6-months follow-up
  Self-reported engagement in PCS / GCS intervention in the different groups.
Validated abstinence and self-reported of PCS-3 vs. GCS-3 | 3- and 6-months follow-up
  Among non-responders to the initial treatments (PCS vs. GCS), compare the two augments treatments: MOS and PCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng X, Song C, Liu K, Zhao S, Yang H, Wang MP. Mobile Phone-Based Smoking-Cessation Intervention in Patients With Chronic Diseases in China: A Sequential Multiple Assignment Randomized Trial. Nicotine Tob Res. 2025 Feb 24;27(3):502-510. doi: 10.1093/ntr/ntae230. PMID 39324617